CLINICAL TRIAL: NCT06187116
Title: Physiotherapist Led Triage in Primary Care for Patients With Hip or Knee Osteoarthritis
Brief Title: Physiotherapist Led Triage in Primary Care for Patients With Hip or Knee OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PT-triage primary care OA
Record Dates: First submitted 2023-05-22; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Physiotherapist; Orthopaedic triage; Quality of care; Surgery Conversion rate
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist led orthopaedic triage (Experimental): Patients who are randomised to PT led triage will be scheduled for a consultation with a physiotherapist (PT) at a rehabilitation clinic in primary care in the Region Västra Götaland.
  Interventions: Other: Physiotherapist consultation
- Usual care (Active Comparator): Patients who are randomised to usual care will be sceduled according to standard procedure for an orthopaedic surgeon (OS) consultation at the orthopaedic department of a hospital in the Region Västra Götaland.
  Interventions: Other: Orthopaedic surgeon consultation

INTERVENTIONS:
Other: Physiotherapist consultation — The consultation with the PT is 40-45 minutes long according to usual care and includes patient history, assessment and management according to an assessment template. If the patient is found not to be appropriate for surgery they can receive the following; 1) self-care without follow up appointment, 2) referral to PT in primary care for rehabilitation, 3) referral back to general practitioner (GP) for new tests/assessments/medication. If the patient is found to be appropriate for surgery, and wishes to undergo surgery, or if the PT in the study wants a second opinion, the patient is 4) referred for orthopaedic consultation for surgical consideration.
  Arms: Physiotherapist led orthopaedic triage
Other: Orthopaedic surgeon consultation — The consultation with the OS is 20-30 minutes long and includes medical history, assessment and management plan, all according to usual care. It the patient is found not to be appropriate for surgery they can receive the following; 1) self-care without follow up appointment, 2) referral to PT in primary care for rehabilitation, 3) referral back to GP for new tests/assessments/medication. If the patient is found appropriate for surgery, and wishes to undergo surgery, the patient is 4) scheduled for surgery.
  Arms: Usual care

SUMMARY:
The overall aim with the study is to evaluate physiotherapist led triage in primary care compared to usual care (assessment by an orthopaedic surgeon in an orthopaedic department) for patients with hip or knee osteoarthritis referred for orthopaedic consultation.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate if there is any difference in perceived quality of care using the item "I received the best possible examination and treatment (as far as I can tell)" between physiotherapist led (PT led) triage in primary care compared to usual care (assessment by an orthopaedic surgeon (OS) in an orthopaedic department) for patients with hip or knee osteoarthritis (OA) referred for orthopaedic consultation. Furthermore, to evaluate whether there is any difference in 2) perceived quality of care as a whole, 3) management outcome and hip/knee replacement surgery conversion rate, 4) patient reported outcome measures such as health related quality, pain and function in short and long term and 5) costs between the two care models.

ELIGIBILITY:
Patients with hip or knee OA assessed by a GP at any of the included health care centers in the study, and referred on for orthopaedic consultation to any of the included hospitals in the Västra Götaland.

Inclusion Criteria:

* primary OA in hip or knee
* understands and speak Swedish

Exclusion Criteria (if stated in the referral)

* Previously been assessed for the same condition by an orthopaedic surgeon
* Referred by an orthopaedic surgeon
* Secondary OA due to fractures or osteonecrosis of the femoral head
* Referral to a specific orthopaedic surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
"I received the best possible examination and treatment (as far as I can tell)" | Within a week after assessment
  One item from the questionnaire Quality from the Patients Perspective (QPP). The patients rate how they perceive the quality of care on a 4-point Likert scale ranging from 1 (do not agree at all) to 4 (completely agree).
  This item was chosen as main outcome since it was found the be representative of quality of care, and as it assess the desired outcome, by the subjective judgement of experts in the field (five physiotherapists and one orthopaedic surgeon).

SECONDARY OUTCOMES:
Quality from the Patients Perspective (QPP) | Within a week after assessment
  Patient perception of the care quality as a whole using the questionnaire Quality from the Patient Perspective (QPP). A valid and reliable measure of patients' perception of quality of care regarding four dimensions: caregivers' medical-technical competence; care organizations' physical-technical conditions; degree of identity-orientation in the caregivers' attitudes and actions; and the care organizations' socio-cultural atmosphere. Each item is evaluated in two ways using a 4-point Likert scale; first the patients rate how they perceive the quality of care ranging from 1 (do not agree at all) to 4 (completely agree). The patients then rate how important that aspect of care is ranging from 1 (little or no importance) to 4 (of the very highest importance). Each item also has a "not applicable" response option.
Waiting times | 12 months after the assessment
  Waiting time from the day of referral to the day of assessment for assessment with PT and OS respectively, measured in days.
Management outcome incl Surgery Conversion Rate (SCR) | 12 months after the assessment
  The number of patients who receive; advice on self-care without follow up appointment (1), referral to physiotherapist in primary care for rehabilitation (2), referral back to the GP (3) or (4) referral for orthopaedic surgery and Surgery Conversion Rate (The number of patients referred for orthopaedic consultation compared with the number of patients who were appropriate for surgery).
EuroQol 5 D (EQ-5D-5L) | Baseline
  Patient reported Quality of life will be measured using the EuroQol 5 D (EQ-5D-5L), a valid and reliable measure of health-related quality of life and consists of 5 items. General health is measured using a VAS scale (0 to 100) with 100 being the best possible health state.
EuroQol 5 D (EQ-5D-5L) | Change from baseline to three months after assessment
  Patient reported Quality of life will be measured using the EuroQol 5 D (EQ-5D-5L), a valid and reliable measure of health-related quality of life and consists of 5 items. General health is measured using a VAS scale (0 to 100) with 100 being the best possible health state.
EuroQol 5 D (EQ-5D-5L) | Change from baseline to 12 months after assessment
  Patient reported Quality of life will be measured using the EuroQol 5 D (EQ-5D-5L), a valid and reliable measure of health-related quality of life and consists of 5 items. General health is measured using a VAS scale (0 to 100) with 100 being the best possible health state.
Forgotten Joint Score (FJS) | Baseline
  Patient reported pain and function will be measured using the Forgotten Joint Score (FJS), a valid and reliable questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a high score is better.
Forgotten Joint Score (FJS) | Change from baseline to three months after assessment
  Patient reported pain and function will be measured using the Forgotten Joint Score (FJS), a valid and reliable questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a high score is better.
Forgotten Joint Score (FJS) | Change from baseline to 12 months after assessment
  Patient reported pain and function will be measured using the Forgotten Joint Score (FJS), a valid and reliable questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a high score is better.
Hip / Knee injury and Osteoarthritis Outcome Score (HOOS-12/KOOS-12) | Baseline
  Patient reported pain and function will be measured using the The 12-item short form of the Hip / Knee injury and Osteoarthritis Outcome Score (HOOS-12/KOOS-12), a valid and reliable short form questionnaires with 12 of the 42-item HOOS/KOOS that provides pain, function and quality of life scale scores and a summary hip/knee impact score. Each item is graded on a 5-point likert scale as well as a summated score graded from 0 to 100, with 100 being the best possible score.
Hip / Knee injury and Osteoarthritis Outcome Score (HOOS-12/KOOS-12) | Change from baseline to three months after assessment
  Patient reported pain and function will be measured using the The 12-item short form of the Hip / Knee injury and Osteoarthritis Outcome Score (HOOS-12/KOOS-12), a valid and reliable short form questionnaires with 12 of the 42-item HOOS/KOOS that provides pain, function and quality of life scale scores and a summary hip/knee impact score. Each item is graded on a 5-point likert scale as well as a summated score graded from 0 to 100, with 100 being the best possible score.
Hip / Knee injury and Osteoarthritis Outcome Score (HOOS-12/KOOS-12) | Change from baseline to 12 months after assessment
  Patient reported pain and function will be measured using the The 12-item short form of the Hip / Knee injury and Osteoarthritis Outcome Score (HOOS-12/KOOS-12), a valid and reliable short form questionnaires with 12 of the 42-item HOOS/KOOS that provides pain, function and quality of life scale scores and a summary hip/knee impact score. Each item is graded on a 5-point likert scale as well as a summated score graded from 0 to 100, with 100 being the best possible score.
Costs | Within 24 months after assessment
  Healthcare consumption (such as visits, further investigations, surgical costs) in primary and secondary healthcare in connection to the patients hip/knee osteoarthritis will be collected from the Swedish Västra Götaland database VEGA. Standard costs for primary care visits will be used to analyse costs. Costs per patient for secondary care will be collected from the Västra Götaland Region database KPP. Sick leave costs will be collected from the Swedish Social Insurance Agency.

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Time Frame: Data will become available upon reasonable request after publication of results
Access Criteria: Analyses and additional data will be available upon reasonable request